CLINICAL TRIAL: NCT00880165
Title: Cost Effective Strategy to Evaluate Veterans With Sleep Apnea
Brief Title: Cost Effectiveness of Ambulatory Management for Veterans With Sleep Apnea
Acronym: VSATT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IIR 04-021
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: Polysomnogram; Continuous positive airway pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): In-laboratory testing followed by continuous positive airway pressure treatment
  Interventions: Device: Continuous positive airway pressure apparatus
- Arm 2 (Active Comparator): Home unattended testing followed by continuous positive airway pressure treatment
  Interventions: Device: Continuous positive airway pressure apparatus

INTERVENTIONS:
Device: Continuous positive airway pressure apparatus — Veterans randomized to both arms who are diagnosed with obstructive sleep apnea will be started on treatment with continuous positive airway pressure.
  Other Names: CPAP

SUMMARY:
This research study is comparing home and in-laboratory testing of veterans with suspected obstructive sleep apnea, a common breathing disorder during sleep. It is hoped that home testing will be equally effective in improving quality of life but have lower cost than in-lab testing. These findings will allow veterans to have greater access to diagnosis and treatment of their sleep apnea.

DETAILED DESCRIPTION:
Objective: The overall goal of the project is to improve access to care for veterans with suspected obstructive sleep apnea (OSA), a breathing disorder during sleep characterized by repetitive closure of the pharyngeal airway. Portable monitors are commercially available to diagnose participants with suspected OSA and establish the continuous positive airway pressure (CPAP) setting needed for treatment. Their application to home testing is not widely accepted because it is not known whether home testing, when compared to conventional in-lab polysomnograms, is cost effective and produces similar outcomes with regard to participant adherence to CPAP treatment and improvements in functional impairment. The specific goals of the proposed research are to address these barriers by comparing the functional impact, cost, and cost-effectiveness of evaluating veterans with suspected OSA using home versus in-lab testing.

Research Design: In this prospective randomized control trial of equivalency, participants referred to the Philadelphia and Pittsburgh VA Medical Centers for evaluation for OSA will be randomized to either exclusively in-lab or home testing following baseline assessment.

Methodology: In-lab polysomnograms will be performed to diagnose OSA and titrate the pressure setting for subsequent CPAP therapy. Self-administered home testing will consist of an overnight unattended sleep study followed by a 1-week autoCPAP titration trial. Objectively assessed CPAP adherence and its consequent effects on subjective and objective daytime sleepiness, disease specific and general functional impairment, and participant preference will be obtained at 1- and 3-months after starting CPAP treatment and 3-monthly thereafter to the end of study follow-up. Medical service use and cost will be collected for the entire observation period.

Aim 1 will determine if participants with suspected OSA who receive home testing have the same adherence to subsequent CPAP treatment and the same functional outcomes as participants receiving in-lab testing. Primary outcome measures will be 1) objectively measured adherence to CPAP treatment and 2) the global score on the Functional Outcomes of Sleep Questionnaire (FOSQ) to assess the consequent effects of adherence on disease specific functional impairment. Secondary functional outcome measures will assess subjective (Epworth Sleepiness Scale) and objective (Psychomotor Vigilance Test) daytime sleepiness, and general quality of life (SF-12). Hypothesis 1: Despite differences between in-lab versus home testing in terms of technology, time participants interact with health care professionals, and environment, there is no clinically significant decline in mean CPAP adherence and no clinically significant reduction in functional outcomes in participants receiving home versus in-lab testing.

Aim 2 will compare the differences in cost and quality-adjusted life years saved (QALYS) between home versus in-lab testing to estimate a cost-effectiveness ratio. Participant preference will be assessed with the EuroQol (EQ-5D) and Health Utilities Index 2 (HUI). Hypothesis 2a: Average total health-care delivery cost is lower for veterans receiving home testing relative to those receiving in-lab testing. Hypothesis 2b: Because we believe that at-home testing will have lower costs and equivalent outcomes, we will be 90% confident that the cost per QALY ratio comparing at-home testing with in-lab testing will be less than $100,000.

Clinical Relationship: We need to determine the most cost effective way to diagnose veterans with OSA and initiate them on CPAP treatment. If the results show that home testing produces clinical outcomes that are not significantly clinically inferior and similar or reduced costs compared with in-lab testing, decision makers can be confident that home monitors can be used to diagnose and treat OSA and that improving veterans' access to care for OSA need not require construction of additional, costly sleep labs.

Findings: We anticipate that the results of Aim 1 will demonstrate that participants receiving in-lab versus home testing have similar clinical outcomes. We further anticipate that Aim 2 will demonstrate that home testing is more cost effective than in-lab testing. If confirmed, these findings will lead to wide acceptance of home portable monitor testing and increase veteran access to care.

ELIGIBILITY:
Inclusion Criteria:

Individuals willing to participate must meet the following eligibility criteria prior to enrollment:

* Patients referred for a sleep evaluation for suspected sleep apnea.
* Age 18 years or older
* Living within 90 miles of the Sleep Center.

Exclusion Criteria:

Individuals will be excluded from the study for the following reasons:

* Unable or unwilling to provide informed written consent.
* Lack of telephone access or inability to return for follow-up testing.
* A history of prior sleep evaluations, OSA treatment, or sleep disorder in addition to OSA.
* A clinically unstable chronic medical condition as defined by a new diagnosis or change in medical management in the previous 3 months of cardiac disease, thyroid disease, diabetes, depression or psychosis, cirrhosis, or recently diagnosed cancer.
* Individuals already on long term oxygen therapy or requiring bilevel positive airway pressure.
* Individuals with rotating shift work or irregular work schedules over the last 6 months.
* Suspected or confirmed to be pregnant. A pregnancy test will be performed using the urine sample obtained at the initial visit.
* Inability to complete the Assessment Battery - e.g. less than a 5th grade reading level

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2006-11; Primary Completion 2009-07 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel T. Kuna, MD, Principal Investigator — VA Medical Center, Philadelphia
Locations (2):
- United States (2):
  - Leonard Davis Institute of Health Economics, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Sunwoo B, Kuna ST. Ambulatory management of patients with sleep apnea: is there a place for portable monitor testing? Clin Chest Med. 2010 Jun;31(2):299-308. doi: 10.1016/j.ccm.2010.02.003. PMID 20488288
- [Result] Kuna ST, Gurubhagavatula I, Maislin G, Hin S, Hartwig KC, McCloskey S, Hachadoorian R, Hurley S, Gupta R, Staley B, Atwood CW. Noninferiority of functional outcome in ambulatory management of obstructive sleep apnea. Am J Respir Crit Care Med. 2011 May 1;183(9):1238-44. doi: 10.1164/rccm.201011-1770OC. Epub 2011 Jan 21. PMID 21471093

RESULTS

PARTICIPANT FLOW:
Groups:
- In-laboratory Testing: In-laboratory testing
  Continuous positive airway pressure apparatus: Veterans randomized to both arms who are diagnosed with obstructive sleep apnea will be prescribed continuous positive airway pressure treatment.
- Home Unattended Testing: Home unattended testing
  Continuous positive airway pressure apparatus: Veterans randomized to both arms who are diagnosed with obstructive sleep apnea will be prescribed continuous positive airway pressure treatment.
Period: Overall Study
Arm/Group | In-laboratory Testing | Home Unattended Testing
Started | 148 | 148
Completed | 86 | 98
Not Completed | 62 | 50
Not completed — Withdrawal by Subject | 27 | 23
Not completed — Not diagnosed with OSA | 14 | 8
Not completed — Required BIPAP or oxygen treatment | 12 | 4
Not completed — Lost to follow | 9 | 15

BASELINE CHARACTERISTICS:
Population: Veterans referred to the participating sleep centers for evaluation of obstructive sleep apnea
Groups:
- Arm 1: In-laboratory testing
  Continuous positive airway pressure apparatus: Veterans randomized to both arms who are diagnosed with obstructive sleep apnea will be started on treatment with continuous positive airway pressure.
- Arm 2: Home unattended testing
  Continuous positive airway pressure apparatus: Veterans randomized to both arms who are diagnosed with obstructive sleep apnea will be started on treatment with continuous positive airway pressure.
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 148 | 148 | 296
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (10.4) | 55.1 (10.3) | 53.2 (10.4)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 137 | 135 | 272
  >=65 years | 11 | 13 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 138 | 135 | 273
Region of Enrollment [Number; unit: participants]
  United States | 148 | 148 | 296
Functional Outcome of Sleep Questionnaire [Mean (Standard Deviation); unit: units on a scale] — Self-administered validated questionnaire assessing functional outcomes in patients with obstructive sleep apnea. The FOSQ total score range is from 1 to 20 with higher scores indicating better functional outcome. The FOSQ has 5 subscale scores: activity level, vigilance, intimacy and sexual relationships, general productivity, social outcome, The range of subscale scores is from 1 to 4 with higher scores indicating better function. The total score is calculated as the mean of the subscales multiplied by 5.
  units on a scale | 14.7 (2.9) | 15.0 (3.2) | 14.9 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: Cost
Description: VA sleep-study and treatment medical service use will be derived from the case report form; and costed out using VA acquisition costs. Other medical service use will be derived from VA administrative records. Non-VA medical service use will be derived from patient interview and will be costed out using federal reimbursement schedules. Costs will be stratified by whether or not they are related to the diagnosis and treatment of OSA.Cost and preferences are assessed for each entire arm.
Time Frame: Medical service use and cost will be collected every 3 months for the entire observation period. Thus the shortest duration of follow-up in the study is anticipated to be 3 months, while the longest will be 2.25 years.
Population: Participants diagnosed with obstructive sleep apnea who were prescribed continuous positive airway pressure (CPAP) treatment. Of the 148 individuals randomized to each arm, 110 in the in-lab testing arm and 113 in the home testing arm were prescribed CPAP. Results from these 223 subjects were used in the per protocol analysis.
Measure: Number; unit: dollars
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 110 | 113
dollars | 4621 (2) | 4057

2. Secondary Outcome: Functional Outcome of Sleep Questionnaire
Description: Change score from baseline of self-administered validate questionnaire of functional outcome following 3 months of positive airway pressure treatment
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 110 | 113
units on a scale | 1.85 (2.46) | 1.74 (2.81)

3. Secondary Outcome: Continuous Positive Airway Pressure Adherence
Description: Mean daily hours of use of continuous positive airway pressure over the 3 month intervention
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 110 | 113
hours per day | 2.92 (2.32) | 3.49 (2.45)

ADVERSE EVENTS:
Time Frame: Adverse events were collected every 3 months for the entire observation period. Collection of adverse events occurred over 2.25 years in the first enrolled participant and over 3 months in the last enrolled participant.
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/148 | 0/148
Other Adverse Events (participants affected / at risk) | 0/148 | 0/148

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes